CLINICAL TRIAL: NCT03020082
Title: A Multi-centered, Open Label, Phase III Study on Efficacy, Safety of Ritonavir-boosted ASC08 (Danoprevir) in Combination With Peg-IFN and RBV in Treatment-Naive Non-Cirrhotic Patients Who Have Chronic Hepatitis Genotype 1
Brief Title: Efficacy and Safety of Danoprevir/r + PR 12week Triple Therapy in Treatment Naive Non-Cirrhotic G1 CHC China III
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ascletis Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Ascletis Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASC08201503
Record Dates: First submitted 2017-01-05; First posted 2017-01-13 (Estimated); Results first posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2017-01

CONDITIONS: Chronic Hepatitis C
Keywords: Danoprevir; non-cirrhotic; Chinese HCV G1; SVR12
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — danoprevir; Ritonavir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Danoprevir, Ritonavir, Peg-IFN,RBV (Experimental): Participants will receive Ritonavir- boosted Danoprevir 100mg/100mg BID in combination with subcutaneous injection of weekly peginterferon alfa-2a at 180 mcg and RBV administered orally 500mg (5 tablets)( body weight <75Kg) BID, 600mg (6 tablets) BID body weight ≥75Kg for 12 weeks.
  Interventions: Drug: Danoprevir; Drug: Ritonavir; Drug: peginterferon alfa-2a; Drug: RBV

INTERVENTIONS:
Drug: Danoprevir — Danoprevir (DNV)administered orally 100mg BID for 12 weeks;
  Other Names: ASC08
Drug: Ritonavir — Ritonavir administered orally 100mg BID for 12 weeks;
Drug: peginterferon alfa-2a — PEG-IFN abdominal or thigh subcutaneous injection, 180μg, once a week for 12 weeks;
  Other Names: Peg-IFN
Drug: RBV — RBV administered orally 500mg (5 tablets)( body weight <75Kg) BID, 600mg (6 tablets) BID body weight ≥75Kg, for 12 weeks.
  Other Names: Ribasphere®

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Ritonavir-boosted ASC08 (Danoprevir) in Combination with Peg-IFN and RBV in Treatment-Naive Non-Cirrhotic Patients Who Have Chronic Hepatitis Genotype 1.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* Chronic HCV infection (≥ 6 months)
* Serum HCV RNA of ≥ 1 × 104 IU/mL are documented
* Hepatitis C virus GT1
* Never received prior-treatment for HCV with interferon, RBV, or other direct-acting or host-targeting antivirals for HCV
* Non-cirrhosis patients: Non-cirrhosis is defined (1)Fibroscan defined as: ˂ 14.6 kPa during screening period, or liver biopsy determined 1 year before recruiting (Metavir score ˂ 3);(2) during screening period 9.6<Fibroscan indicator ≤12.9, liver biopsy need to confirm non-cirrhosis.
* Others as specified in the detailed protocol

Exclusion Criteria:

* Patients with Fibroscan detection value > 12.9 kPa, or histologic examination for liver cirrhosis patients
* Presence or history of non-hepatitis C chronic liver disease (e.g. HH, AIH, Wilson's disease, α1 antitrypsin deficiency, drug- or toxin-induced liver disease)
* History of liver cell cancer, or suspected hepatocellular carcinoma (HCC) patients before or during screening , or imaging studies found suspicious nodules, or AFP > 50 ng/mL
* Positive hepatitis A antibody，positive hepatitis B surface antigen，HIV antibody
* Presence or history of nervous system diseases and/or mental illness, inability to control oneself or express oneself.
* Patients with obvious cardiovascular dysfunction
* Pregnant or nursing female, nor unwilling to take reliable contraception
* Others as specified in the detailed protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2016-06; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Huoling Tang, PhD, Study Director — Ascletis Pharmaceuticals Co., Ltd.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wei L, Shang J, Ma Y, Xu X, Huang Y, Guan Y, Duan Z, Zhang W, Gao Z, Zhang M, Li J, Jia J, Yang Y, Wen X, Wang M, Jia Z, Ning B, Chen Y, Qi Y, Du J, Jiang J, Tong L, Xie Y, Wu JJ. Efficacy and Safety of 12-week Interferon-based Danoprevir Regimen in Patients with Genotype 1 Chronic Hepatitis C. J Clin Transl Hepatol. 2019 Sep 28;7(3):221-225. doi: 10.14218/JCTH.2019.00018. Epub 2019 Jul 22. PMID 31608213

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Danoprevir, Ritonavir, Peg-IFN,RBV
Started | 141
Completed | 138
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Danoprevir, Ritonavir, Peg-IFN,RBV
Number analyzed (Participants) | 141
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70
  Male | 71
Race (NIH/OMB) [Count of Participants; unit: Participants] — Asia
  Participants
    American Indian or Alaska Native | 0
    Asian | 141
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 0
    More than one race | 0
    Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Sustained Virologic Response 12 Weeks After Discontinuation of Therapy (SVR12)
Time Frame: 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Danoprevir, Ritonavir, Peg-IFN,RBV
Number analyzed (Participants) | 141
Participants | 136

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Danoprevir, Ritonavir, Peg-IFN,RBV
All-Cause Mortality (participants affected / at risk) | 0/141
Serious Adverse Events (participants affected / at risk) | 5/141
Other Adverse Events (participants affected / at risk) | 76/141
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Danoprevir, Ritonavir, Peg-IFN,RBV (N=141)
neutropenia (Blood and lymphatic system disorders) | 1
Ventricular tachyarrhythmia (Cardiac disorders) | 1
Tuberculosis (Infections and infestations) | 1
Transient ischemic attack (Metabolism and nutrition disorders) | 1
Acquired digital fibrokeratoma (Eye disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Danoprevir, Ritonavir, Peg-IFN,RBV (N=141)
Anemia (Blood and lymphatic system disorders) | 76
Fever (Infections and infestations) | 53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Ascletis, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met: The study has been completed at all study sites for at least 3 years.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-03-21): https://cdn.clinicaltrials.gov/large-docs/82/NCT03020082/SAP_000.pdf
  • Study Protocol (2017-01-16): https://cdn.clinicaltrials.gov/large-docs/82/NCT03020082/Prot_001.pdf